CLINICAL TRIAL: NCT02056041
Title: Selection Criteria for Safe Hepatectomy for Hepatocellular Carcinoma: Validation on 336 Consecutive Hepatectomies.
Brief Title: Selection Criteria for Safe Hepatectomy for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Other Study IDs: SafeSurgeryHCC
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Hepatectomy; Hepatecellular Carcinoma; Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hepatectomy for HCC: Patients submitted to surgery for HCC
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy
  Other Names: Liver surgery; Liver resection; Hepatic resection

SUMMARY:
Selection criteria for safe hepatectomy for HCC are not well established. The aim of this study was the validation of the selection criteria for safe hepatectomy for hepatocellular carcinoma.

DETAILED DESCRIPTION:
All consecutive patients submitted to hepatectomy for HCC based on the same preoperative selection criteria from our prospectively-maintained liver unit database. Such criteria included the value of bilirubin (BIL), the value of cholinesterases (CHE), the presence of ascites, the presence of esophageal varices, and the rate of residual liver volume.

ELIGIBILITY:
Inclusion Criteria:

* any patient with HCC submitted to hepatic resection at our Unit in the established frame time

Exclusion Criteria:

* any patient with missing data or lost at follow-up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The records of 336 consecutive patients who were submitted to hepatectomy between 2004-2012 were reviewed.
Sampling Method: Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2004-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety of surgery for HCC | 90 days
  The primary endpoint was the validation of our selection criteria for safe hepatectomy for HCC in regards to postoperative complications. The role of total bilirubin and cholinesterases was analzyed together with other clinical parameters.

SECONDARY OUTCOMES:
Score systems HCC | 90 days
  The secondary endpoint was the testing of the most common score systems for HCC, which are the CPT score, the MELD score, and the APRI score.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Derived] Donadon M, Costa G, Cimino M, Procopio F, Fabbro DD, Palmisano A, Torzilli G. Safe hepatectomy selection criteria for hepatocellular carcinoma patients: a validation of 336 consecutive hepatectomies. The BILCHE score. World J Surg. 2015 Jan;39(1):237-43. doi: 10.1007/s00268-014-2786-6. PMID 25217112